CLINICAL TRIAL: NCT01274455
Title: PILOT STUDY OF GENE THERAPY FOR LOCALLY ADVANCED PANCREATIC ADENOCARCINOMA WITH INTRATUMOURAL INJECTION OF JetPEI/DNA COMPLEXES WITH ANTITUMOURAL EFFECT AND CHEMOSENSITIZING ACTIVITY FOR GEMCITABINE
Brief Title: Gene Therapy of Pancreatic Ductal Adenocarcinoma
Acronym: TherGAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Clinical Research Center, Toulouse (Other); CAYLA-INVIVOGEN (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0401401
Record Dates: First submitted 2010-12-10; First posted 2011-01-11 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Gene therapy; pancreatic carcinoma; gemcitabine; endoscopic ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapy (Experimental)
  Interventions: Genetic: Gene Therapy product CYL-02 = plasmid DNA pre-complexed to linear polyethylenimine encoding sst2 + dck::umk genes

INTERVENTIONS:
Genetic: Gene Therapy product CYL-02 = plasmid DNA pre-complexed to linear polyethylenimine encoding sst2 + dck::umk genes — Intratumoral injection of the gene therapy product CYL-02 (2,5 ml within the primary tumor under endoscopic ultrasound guidance an under propofol anaesthesia). The intratumor injection of CYL-02 is followed by three IV infusions of Gemcitabine (1000 mg/m2) at 48 hours and then every two weeks. A second Intratumoral injection of the gene therapy product CYL-02 is performed at a same dosage and volume 30 days after the first administration followed by Three infusions of gemcitabine (1000 mg/m2) according the same rhythm (48 hours and every week) and dose.

SUMMARY:
Near 85% of patients with pancreatic adenocarcinoma are diagnosed with a locally advanced and/or metastatic unresectable tumor. In these patients chemotherapy (such as gemcitabine) is given as a palliative therapy. Aim of the present study is to evaluate the feasibility, tolerance and antitumor effect of repeated intratumoral injection of a gene therapy product (with antitumor and chemo sensitizing effects) combined with gemcitabine in patients with unresectable pancreatic carcinoma.

DETAILED DESCRIPTION:
This is a gene therapy open non randomized phase I trial for advanced and/or metastatic pancreatic cancer patients. The protocol is based on the administration of increasing doses of a plasmid DNA pre-complexed to PEI (polyethylenimine - non-viral vector) that encodes two genes (somatostatin receptor subtype 2 named sst2 and deoxycitidine kinase :: uridylmonophosphate kinase named dck::umk) which exhibit complementary therapeutic effects. Both transgenes induce an antitumor bystander effect and render gemcitabine treatment more efficient. Intratumor injections of the gene therapy product (CYL-02) will be performed by transgastric or transduodenal route under endoscopic ultrasound guidance. Each injection will be followed standard gemcitabine IV administration every week (1000 mg/m2). Two intratumor injections of a same dose of CYL-02 will be administered at one month interval. Four increasing doses (125 µg, 250 µg, 500 µg and 1 mg) will be tested by group of 6 patients. The primary objectives are: evaluation of local pancreatic and general tolerance; the secondary objectives are: possible tumor volume regression, secondary respectability, evaluation of transgene biodistribution.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a pancreatic adenocarcinoma histologically proven and/or a solid pancreatic mass associated with on or multiple metastatis from pancreatic origin (histologically proven)
* Patient with a non resectable pancreatic adenocarcinoma (on preoperative CT-scan and/or endoscopic ultrasound evaluation)
* Pancreatic tumor that could be evaluated by endoscopic ultrasound (no digestive stenosis, no gastrectomy)
* Patient with no contraindication to général anaesthesia.
* Karnofsky index >= 70%
* Written informed consent given

Exclusion Criteria:

* - Exclusion period for another clinical trial or research protocol.
* Patient unable to read or understand information/consent formula or unable to decide alone for his participation to the trial
* Patient under tutelage
* Pregnant woman or able to procreate without contraception.
* Patient with pancreatic cystic tumor or pancreatic pseudocyst.
* Patient with pancreatic tumor different from adenocarcinoma (endocrine, metastasis).
* Patient contraindication to Gemzar® :

  * Hypersensitivity to Gemcitabine.
  * Decision of radiotherapy
  * Granulocytes < 1000/mm3
  * Thrombocytes < 100 000/mm3
* Patient not efficiently treated for jaundice (biliary stent or bypass) if present at time of diagnosis
* Contraindication for fine needle aspiration biopsy under endoscopic ultrasound (hemostasis trouble).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Feasability and security : Number of Participants with Adverse Events | 60 days
  Feasibility, security (pancreas and general) of intratumor injections of the gene therapy product (CYL-02 plasmid DNA pre-complexed to PEI encoding sst2 dck::umk) administered under endoscopic ultrasound guidance and followed by gemcitabine treatment at standard doses.

SECONDARY OUTCOMES:
Antitumoral effect: secondary resecability, transgenes diffusion | 60 days
  antitumoral effect, secondary resecability, transgenes diffusion (urine and blood) and expression (tumor).

CONTACTS AND LOCATIONS:
Overall Officials: Louis BUSCAIL, MD,PhD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- Toulouse Universitary Hospital (Rangueil), Department of Gastroenterology At Rangueil Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No